CLINICAL TRIAL: NCT05379647
Title: QN-019a as a Monotherapy and in Combination With Anti-CD20 Monoclonal Antibodies in Subjects With B-Cell Malignancies
Brief Title: Natural Killer (NK) Cell Therapy for B-Cell Malignancies
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Collaborators: Hangzhou Qihan Biotech Co., Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Clinical Professor, Zhejiang University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-002 (QN-019a)
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: B-cell Lymphoma; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma | interventions — Rituximab; Cyclophosphamide; fludarabine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QN-019a in Combination with Monoclonal Antibodies (Experimental): QN-019a in Combination with Rituximab in adult subjects with r/r B-cell lymphoma.
  Interventions: Drug: QN-019a; Drug: Rituximab; Drug: Cyclophosphamid; Drug: Fludarabine; Drug: VP-16
- QN-019a Monotherapy (Experimental): QN-019a Monotherapy in adult subjects with r/r B-ALL
  Interventions: Drug: QN-019a; Drug: Cyclophosphamid; Drug: Fludarabine; Drug: VP-16

INTERVENTIONS:
Drug: QN-019a — Experimental Interventional Therapy
Drug: Rituximab — Monoclonal Antibody
  Arms: QN-019a in Combination with Monoclonal Antibodies
Drug: Cyclophosphamid — Lympho-conditioning Agent
Drug: Fludarabine — Lympho-conditioning Agent
Drug: VP-16 — Lympho-conditioning Agent

SUMMARY:
This is an open-label, Phase I study of QN-019a (allogeneic CAR-NK cells targeting CD19) as monotherapy in relapsed/refractory B-cell Acute Lymphoblastic Leukemia (B-ALL) and in combination with Rituximab in relapsed/refractory B-cell Lymphoma.

This clinical study is to evaluate the safety, tolerability and preliminary efficacy of QN-019a in patients with relapsed/refractory B-cell lymphoma or B-ALL. Up to 22-36 patients will be enrolled.

DETAILED DESCRIPTION:
This is an open-label, Phase I study of QN-019a (allogeneic CAR-NK cells targeting CD19) as monotherapy in relapsed/refractory B-cell Acute Lymphoblastic Leukemia (B-ALL) and in combination with Rituximab in relapsed/refractory B-cell Lymphoma.

This clinical study is to evaluate the safety, tolerability and preliminary efficacy of QN-019a in patients with relapsed/refractory B-cell lymphoma or B-ALL, where a "3+3" enrollment schema will be utilized at dose escalation stage. Up to 24-36 patients will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of B-cell lymphoma or B-ALL as described below:

B-cell Lymphoma:

* Histologically documented lymphomas expected to express CD19 and CD20
* Relapsed/refractory disease following at least two prior systemic treatment regimens, or relapsed after the autologous hematopoietic stem cell transplantation (HSCT)

B-ALL:

* Diagnosis of B-ALL that expected to express CD19
* Relapsed/refractory disease following prior systemic treatment regimens

ALL SUBJECTS:

* Provision of signed and dated informed consent form (ICF)
* Age ≥ 18 years old
* Stated willingness to comply with study procedures and duration
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function as defined in the protocol
* Donor specific antibody (DSA) to QN-019a: MFI <= 2000
* At least 3 weeks after the last systemic immunochemotherapy treatment
* The estimated survival days are expected to be over 3 months

Key Exclusion Criteria:

ALL SUBJECTS:

* Females who are pregnant or lactating
* Evidence of insufficient organ function as defined in the protocol
* ECOG Performance Status ≥2
* Prior allogeneic hematopoietic stem cell transplant (HSCT) or allogeneic CAR-T/CAR-NK within 6 months of Day 1, or ongoing requirement for systemic GvHD therapy
* Currently receiving or likely to require systemic immunosuppressive therapy
* Known active central nervous system (CNS) involvement by malignancy. Non-malignant CNS disease such as stroke, epilepsy, or neurodegenerative disease
* Clinically significant cardiovascular disease as defined in the protocol
* Known HIV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* Donor specific antibody (DSA) to QN-019a: MFI > 2000
* Other comorbid conditions and concomitant medications prohibited as per study protocol
* Investigator-assessed presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of subjects with Dose Limiting Toxicities within each dose level cohort | Day 28
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Day 28
  Incidence, nature, and severity of treatment related adverse events will be evaluated.

SECONDARY OUTCOMES:
Objective response rate (ORR) of QN-019a as monotherapy in r/r B-ALL and in combination with Rituximab in r/r B-cell Lymphoma | From baseline tumor assessment up to approximately 2 years after last dose of QN-019a
Duration of response (DOR) of QN-019a as monotherapy in r/r B-ALL and in combination with Rituximab in r/r B-cell Lymphoma | Up to approximately 2 years after last dose of QN-019a
Progression-free survival (PFS) of QN-019a in combination with Rituximab in r/r B-cell Lymphoma | Up to approximately 2 years after last dose of QN-019a
Overall survival (OS) of QN-019a as monotherapy in r/r B-ALL and in combination with Rituximab in r/r B-cell Lymphoma | Up to approximately 2 years after last dose of QN-019a
Determination of the pharmacokinetics (PK) of QN-019a cells in peripheral blood | Up to approximately 2 years after last dose of QN-019a
  The PK of QN-019a in peripheral blood will be reported as the relative percentage of product (QN-019a) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points
Event-free survival (EFS) of QN-019a as monotherapy in r/r B-ALL | Up to approximately 2 years after last dose of QN-019a

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PhD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China